CLINICAL TRIAL: NCT00280709
Title: Covered Versus Uncovered Metal Stents for Management of Distal Malignant Biliary Obstruction? Results of a Randomized Prospective Study.
Brief Title: Biliary Metal Stent Study: Metal Stents for Management of Distal Malignant Biliary Obstruction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Eric Kullman, M.D., Associate Professor, Department of Surgery, University Hospital, Linkoping, Sweden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ELLA
Record Dates: First submitted 2006-01-20; First posted 2006-01-23 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2010-12

CONDITIONS: Bile Duct Obstruction; Pancreatic Cancer; Gallbladder Cancer; Bile Duct Cancer
Keywords: Bile duct; Bile duct obstruction; Biliary stent; Metal stent; ERCP; Patency; Complication; Stent occlusion
MeSH Terms: conditions — Cholestasis; Pancreatic Neoplasms; Gallbladder Neoplasms; Bile Duct Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Covered metal stent
  Interventions: Device: "Nitinella" ; SX-ELLA Stent Biliary (biliary metal stent)
- 2 (Active Comparator): Uncovered metal stent
  Interventions: Device: "Nitinella" ; SX-ELLA Stent Biliary (biliary metal stent)

INTERVENTIONS:
Device: "Nitinella" ; SX-ELLA Stent Biliary (biliary metal stent) — Nitinella covered (arm 1) or uncovered (arm 2) biliary metal stent. Maximum diameter 10 mm, length 52 or 72 mm

SUMMARY:
The primary purpose is to compare patency of two different types of biliary metal stents, i.e. covered versus uncovered Nitinella metal stent. Secondary purposes are to determine frequency of complications in the two groups, e.g. cholecystitis, pancreatitis, and cholangitis.

ELIGIBILITY:
Inclusion Criteria:

* 20 years of age or older
* oral and written information given and informed consent obtained
* clinical data in accordance with malignant bile duct obstruction
* ultrasonography signs of extrahepatic malignant common bile duct obstruction
* typical radiological findings at ERCP of malignant common bile duct stenosis
* proximal margin of the bile duct stenosis at least 2 cm from the hepatic confluence
* bilirubin > 50 micromol/L
* radical surgery estimated not possible (temporary stenting with insertion of a plastic stent can be obtained but should be replaced by a metal stent within 4 weeks after the first ERCP procedure, and the patient is randomized at the time of insertion of the metal stent)

Exclusion Criteria:

* patients with active hepatitis or other hepatic diseases that may cause jaundice
* informed consent not obtained
* metastasis with numerous significant intrahepatic stenosis causing blockage of one or more segments of the liver (if no segment blockage, liver metastasis is not an exclusion criteria)
* the patient is probably a candidate for surgical resection
* suspicion of a non-malignant bile duct obstruction, e.g. stones or benign stenosis (should initiate further investigations)
* the proximal end of the stenosis is located within 2 cm from the hepatic confluence
* the patient has previously undergone BII or Roux-en-Y gastric resection, or has a significant duodenal obstruction making ERCP difficult
* previously (more than 4 weeks earlier) treated with a bile duct stent
* severe coagulation disturbance (PK-INR > 1.6)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2006-01; Primary Completion 2008-10 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Clinical follow-up every month, starting one month after stent insertion. Clinical and/or laboratory signs of stent dysfunction? | 12 months after stent insertion

CONTACTS AND LOCATIONS:
Overall Officials: Eric P Kullman, M.D., Study Chair — Department of Surgery, University Hostpital, Linkoping, Sweden.; Claes Soderlund, M.D., Principal Investigator — Department of Surgery, Sodersjukhuset, Stockholm, Sweden.; Bo Ohlin, M.D., Principal Investigator — Department of Surgery, Central Hospital of Blekinge, Karlskrona, Sweden.; Ervin Toth, M.D., Principal Investigator — Department of Endoscopy, University Hospital MAS, Malmö, Sweden.; Carl-Eric Leijonmarck, M.D., Principal Investigator — Department of Surgery, S:t Goran Hospital, Stockholm, Sweden.; Eduard Jonas, M.D., Principal Investigator — Department of Surgery, Danderyd Hospital, Stockholm, Sweden.; Claes Rudberg, M.D., Principal Investigator — Department of Surgery, Central Hospital, Vasteras, Sweden.; Kalev Teder, M.D., Principal Investigator — Department of Surgery, Central Hospital, Norrkoping, Sweden.; Erik Svartholm, M.D., Principal Investigator — Department of Surgery, Ryhov Hospital, Jonkoping, Sweden.; Mehmet Gozen, M.D., Principal Investigator — Department of Surgery, Vastervik Hospital, Vastervik, Sweden.
Locations (1):
- Department of Surgery, University Hospital, Linköping, Sweden

REFERENCES:
- [Derived] Kullman E, Frozanpor F, Soderlund C, Linder S, Sandstrom P, Lindhoff-Larsson A, Toth E, Lindell G, Jonas E, Freedman J, Ljungman M, Rudberg C, Ohlin B, Zacharias R, Leijonmarck CE, Teder K, Ringman A, Persson G, Gozen M, Eriksson O. Covered versus uncovered self-expandable nitinol stents in the palliative treatment of malignant distal biliary obstruction: results from a randomized, multicenter study. Gastrointest Endosc. 2010 Nov;72(5):915-23. doi: 10.1016/j.gie.2010.07.036. PMID 21034892